CLINICAL TRIAL: NCT05923086
Title: A Multi-center, Randomized, Double Blind, Placebo-controlled, Phase 2 Study to Investigate the Efficacy of ORE-001 in Preventing Gastrointestinal Disturbance/ Intolerance in Patients After Longitudinal Laparotomy
Brief Title: Preventing Gastrointestinal Disturbance in Patients After Longitudinal Laparotomy.
Acronym: ORE001PIIPOI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Orexa BV (Industry)
Collaborators: QPS Holdings LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT-2022-503113-31
Record Dates: First submitted 2023-06-09; First posted 2023-06-28 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Ileus Postoperative
Keywords: local anesthetic
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, double blind, placebo-controlled, phase 2 pilot efficacy study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment (4 tablets)
  Interventions: Drug: Placebo
- ORE001 (Experimental): ORE001 treatment (4 tablets)
  Interventions: Drug: ORE001

INTERVENTIONS:
Drug: ORE001 — Administration before major meal
  Other Names: Lidocaine
  Arms: ORE001
Drug: Placebo — Administration before major meal
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled, phase 2 pilot efficacy study.

DETAILED DESCRIPTION:
After assessing eligibility during a screening period (up to 4 weeks before planned surgery), up to 126 female patients are planned to be randomized to one of the two treatment groups.

After the surgery, at POD1 (Post Operative Day 1), all patients will receive the oral study drug (ORE-001 4x 100 mg or 4x placebo) 15-30 minutes before intake of the semi-solid main meal (lunch).

Clinical assessments of efficacy will be conducted based on I-FEED score and VAS (Visual Analogue Scale) abdominal pain score at POD1 to POD8 (or up to POD12 if extended), and the impact of the treatment on the Quality of Life (QoL) of the patients at POD8 (or at POD9 up to POD12 if extended) and at Follow up (FU) in comparison to Baseline values. The impact of the treatment on the QoL will be done by using the specific 36-Item Short Form Survey Instrument (SF-36) QoL questionnaire.

Adverse events (AEs) will be recorded from POD1 to EOS continuously, concomitant medication, and other assessments including vital signs and body weight will be recorded throughout the study (Screening to EOS (End Of Study)).

Urine pregnancy tests (only for females of childbearing potential) will be performed at Screening and Baseline. 12-lead ECG will be performed at Screening, Baseline, POD1 and at Day after last study drug administration.

Safety laboratory assessments on blood (hematology and biochemistry) and urine (routine dip stick test) will be conducted at Screening, Baseline, POD1 and from POD4 every second day until one day after last IMP administration to assess for any changes in the safety endpoints.

Blood albumin will be analyzed on Screening, Baseline, and every POD until one day after last IMP administration to assess for any changes in the safety endpoints.

Interleukin 6 will be analyzed at POD1 and POD6. Patients prematurely terminating the study after administration of at least one dose of the study drug should be subjected to a final examination including safety laboratory assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be able to understand the requirements of the study and give written informed consent prior to study start.
2. Female patients aged between 18 and 75 years (both inclusive).
3. Gynecologic surgery performed completely by longitudinal laparotomy.
4. Patient with ECOG Performance status up to 1.
5. Patient is highly likely to comply with the protocol and complete the study.
6. Patient agrees to be scheduled for peridural catheter (PDC).

Exclusion Criteria:

1. Patient has a history of gastrectomy, total colectomy, stoma creation, short bowel syndrome.
2. Patient has pre-operative ileus.
3. Patient is taking opioid analgesics longer than two post-operative days, exceeding a dosing of 35 mg morphine equivalent per day.
4. Chemotherapy treatment within 10 days after longitudinal surgery.
5. Smoking during the hospital stay.
6. Any contraindication as per summary of product characteristic for the usage of local anesthetics for PDC.
7. History of uncontrolled (at the discretion of the Investigator) cardiovascular, renal and/or hepatic failure.
8. History of severe allergic or anaphylactic reactions, especially to local anesthetics.
9. Clinically significant (at the discretion of the Investigator) deviation from the normal laboratory values.
10. Clinically significant (at the discretion of the Investigator) abnormal ECG.
11. Intake of any class 1B antiarrhythmic drugs if used for antiarrhythmic purpose (e.g., Lidocaine, Mexiletine, Phenytoin) and of any class 3 antiarrhythmic drugs - Kalium channel blockers (e.g., Amiodarone, Dronedarone, Sotalol, Ibutilide, Dofetilide, Bretylium).
12. Significant (at the discretion of the Investigator) symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection (especially with need of antibiotic treatment) within the past 2 weeks prior to study medication administration.
13. Experimental agent within 30 days or ten half-lives, whichever is longer, prior to study medication administration.
14. Pregnancy or planning to become pregnant during the study.
15. Any other condition, which in the opinion of the Investigator precludes the patient's participation in the study.
16. Patients with close affiliation with the Investigator or persons working at the respective study sites or patients who are an employee of the Sponsor.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 126 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
I-FEED Post Operative Day 3 | Post Operative Day 3
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD3. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.

SECONDARY OUTCOMES:
I-FEED Post Operative Day 1 | Post Operative Day 1
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD1. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 2 | Post Operative Day 2
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD2. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 4 | Post Operative Day 4
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD4. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 5 | Post Operative Day 5
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD5. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 6 | Post Operative Day 6
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD6. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 7 | Post Operative Day 7
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD7. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 8 | Post Operative Day 8
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD8. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 9 | Post Operative Day 9
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD9. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 10 | Post Operative Day 10
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD10. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 11 | Post Operative Day 11
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD11. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
I-FEED Post Operative Day 12 | Post Operative Day 12
  To evaluate the efficacy of oral ORE-001 compared to placebo in reducing the gastrointestinal disturbance/intolerance and the occurrence of postoperative ileus (POI) in patients after longitudinal laparotomy defined by scoring of the postoperative I-FEED scores at POD12. The I-FEED score ranges from 0 to 14. The higher the score the more severe are the symptoms.
Number of participants with treatment-related adverse events | Post Operative Day 1-13
  To evaluate the safety and tolerability of oral ORE-001 in comparison to placebo in patients after longitudinal laparotomy at Baseline and up to POD9 (with possible extension to POD13).

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Bonn (UKB)., Bonn
  - Kaiserswerther Diakonie Florence-Nightingale- Krankenhaus, Düsseldorf
  - Klinikum Wolfsburg, Wolfsburg

IPD SHARING:
Plan to Share IPD: No